CLINICAL TRIAL: NCT02471976
Title: Impact of a Computer-assisted Tool to Help Reflection on the Decision to Withhold or to Withdraw Treatments for Surgical Patients in Intensive Care Units
Brief Title: Impact of an Early Palliative Approach
Acronym: LATAREA-IV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: K071203
Record Dates: First submitted 2015-06-01; First posted 2015-06-15 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Criteria of Vulnerability
Keywords: Leonetti law; palliative care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (No Intervention): the centres applies their usual practices
- Group B (Other): strategy promoting early consideration and collegiate vulnerability of patients
  Interventions: Other: strategy promoting early consideration and collegiate vulnerability of patients

INTERVENTIONS:
Other: strategy promoting early consideration and collegiate vulnerability of patients — One day training with the provision of vulnerability criteria inciting an early reflection of the level of therapeutic engagement; sheets available on the internet computer support collegial reflection and traceability of decisions to limit and stop treatments, incorporating the provisions of law known Leonetti
  Arms: Group B

SUMMARY:
Rationale: Medicalized end of life rose profound society questions and debates. Major Laws and scientific society recommendations emerged from those reflections. These texts help withholding/withdrawing life-sustaining treatments allowing a palliative approach and to favor comfort treatments for end of life patients.

Main Objective: To evaluate the impact of a procedure to support reflection on the level of therapeutic involvement for surgical patient (who undergone surgery or not) in ICU after having identified vulnerability criteria early.

Secondary objectives: To assess the usual care of the control group and the impact of the procedure according to ICU type (medical, surgical, mixed); the characteristics of surgical patients concerned by a palliative strategy; the impact of an incentive approach on length of mechanical ventilation and length of stay in the ICU; To measure the extent of information collected concerning the collegial process; the impact of the procedure on caregivers' satisfaction; To count the number of identified conflicts Study type: Prospective, controlled, cluster randomized study of routine care Purpose: Study the implementation of the Act "Leonetti" released on 22 April 2005 calling for a compassionate approach and palliative care for patients at end of life.

Inclusion criteria: Surgical patients (who undergone surgery or not) hospitalized in ICU during the study period Non-inclusion criteria: Patients hospitalized less than 24h; non-surgical patients; patients who don't need ICU care or surveillance; minors; brain-dead patients (at the time of admission) Primary endpoint: Rate of deaths with palliative strategy (withholding or withdrawing treatments) Randomization process: each center is randomized adjusting on type of ICU (medical, surgical, mixed) and number of annual hospitalization volume.

* Control group: ICU usual care
* Intervention group: vulnerability criteria lead to reflection on level of therapeutic involvement, with the help of a written guide.

Number of patients: 2750 surgical patients Number of centers: 45 Study design: usual data will be collected in a secured web-based Case Report Form (CRF) at ICU admission and each time therapeutic strategy will change. Additional data will be collected for the intervention group according to the initial presence or the later apparition of predefined criteria, a standardized reflection procedure will start helped by the implementation of a guide for collegial approach and decision making.

Length: 30 months

ELIGIBILITY:
Inclusion Criteria:

* Surgical patients (who undergone surgery or not) hospitalized in ICU during the study period
* No opposition to the use of data collected from the patient or a relative or inclusion in emergency and non-opposition collected offline

Exclusion Criteria:

* Patients admitted legally dead or brain-dead

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1172 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2014-01 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number of participants dead with palliative strategy | From ICU hospitalization to 6 months after inclusion
  Rate of death with collegial process and withdrawing/withholding treatment

SECONDARY OUTCOMES:
Impact of the procedure according to ICU type | From ICU hospitalization to 6 months after inclusion
Characteristics of surgical patients concerned by a palliative strategy | From ICU hospitalization to 6 months after inclusion
Impact of an incentive approach on length of mechanical ventilation and length of stay in the ICU. | From ICU hospitalization to 6 months after inclusion
Extent of information collected concerning the collegial process | From ICU hospitalization to 6 months after inclusion
Impact of the procedure on caregivers' satisfaction | From ICU hospitalization to 6 months after inclusion
Number of identified conflicts | From ICU hospitalization to 6 months after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Edouard FERRAND, MD, Principal Investigator — Hôpital FOCH
Locations (1):
- Hôpital FOCH, Suresnes, France

REFERENCES:
- [Background] Ferrand E, Jabre P, Vincent-Genod C, Aubry R, Badet M, Badia P, Cariou A, Ellien F, Gounant V, Gil R, Jaber S, Jay S, Paillaud E, Poulain P, Regnier B, Reignier J, Socie G, Tardy B, Lemaire F, Brun-Buisson C, Marty J; French Mort-a-l'Hopital Group. Circumstances of death in hospitalized patients and nurses' perceptions: French multicenter Mort-a-l'Hopital survey. Arch Intern Med. 2008 Apr 28;168(8):867-75. doi: 10.1001/archinte.168.8.867. PMID 18443263
- [Background] Ferrand E, Robert R, Ingrand P, Lemaire F; French LATAREA Group. Withholding and withdrawal of life support in intensive-care units in France: a prospective survey. French LATAREA Group. Lancet. 2001 Jan 6;357(9249):9-14. doi: 10.1016/s0140-6736(00)03564-9. PMID 11197395
- [Background] Ferrand E, Lemaire F, Regnier B, Kuteifan K, Badet M, Asfar P, Jaber S, Chagnon JL, Renault A, Robert R, Pochard F, Herve C, Brun-Buisson C, Duvaldestin P; French RESSENTI Group. Discrepancies between perceptions by physicians and nursing staff of intensive care unit end-of-life decisions. Am J Respir Crit Care Med. 2003 May 15;167(10):1310-5. doi: 10.1164/rccm.200207-752OC. Epub 2003 Jan 24. PMID 12738597
- [Background] Truog RD, Cist AF, Brackett SE, Burns JP, Curley MA, Danis M, DeVita MA, Rosenbaum SH, Rothenberg DM, Sprung CL, Webb SA, Wlody GS, Hurford WE. Recommendations for end-of-life care in the intensive care unit: The Ethics Committee of the Society of Critical Care Medicine. Crit Care Med. 2001 Dec;29(12):2332-48. doi: 10.1097/00003246-200112000-00017. No abstract available. PMID 11801837
- [Background] Ferrand E, Marty J; French LATASAMU Group. Prehospital withholding and withdrawal of life-sustaining treatments. The French LATASAMU survey. Intensive Care Med. 2006 Oct;32(10):1498-505. doi: 10.1007/s00134-006-0292-5. Epub 2006 Aug 2. PMID 16896861
- [Background] Prendergast TJ, Claessens MT, Luce JM. A national survey of end-of-life care for critically ill patients. Am J Respir Crit Care Med. 1998 Oct;158(4):1163-7. doi: 10.1164/ajrccm.158.4.9801108. PMID 9769276
- [Background] Sprung CL, Cohen SL, Sjokvist P, Baras M, Bulow HH, Hovilehto S, Ledoux D, Lippert A, Maia P, Phelan D, Schobersberger W, Wennberg E, Woodcock T; Ethicus Study Group. End-of-life practices in European intensive care units: the Ethicus Study. JAMA. 2003 Aug 13;290(6):790-7. doi: 10.1001/jama.290.6.790. PMID 12915432
- [Background] Ferrand E, Jabre P, Fernandez-Curiel S, Morin F, Vincent-Genod C, Duvaldestin P, Lemaire F, Herve C, Marty J. Participation of French general practitioners in end-of-life decisions for their hospitalised patients. J Med Ethics. 2006 Dec;32(12):683-7. doi: 10.1136/jme.2005.014084. PMID 17145904